CLINICAL TRIAL: NCT04139668
Title: Vivitrol Associated With Behavioural-Relapse Prevention Strategy as Treatment for Cannabis Use Disorder
Brief Title: Vivitrol Treatment for Cannabis Use Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder contract terminated
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 048/2018
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-10

CONDITIONS: Cannabis Use Disorder
MeSH Terms: interventions — Naltrexone; vivitrol; Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vivitrol + MET/CBT (Experimental): All participants will receive three 4ml doses of extended-release naltrexone 380mg (Vivitrol), administered by intramuscular injection. Three injections will be administered to each participant; one injection every 4 weeks for 12 weeks of treatment. In addition, all participants will receive weekly Motivational Enhancement Therapy and Cognitive Behavioral Therapy for 12 weeks.
  Interventions: Drug: Naltrexone 380 MG [Vivitrol]; Behavioral: Motivational Enhancement Therapy and Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Naltrexone 380 MG [Vivitrol] — Three 4ml intramuscular injections of naltrexone 380mg (Vivitrol) administered over 12 weeks (one injection every 4 weeks)
  Other Names: Extended release naltrexone; Injectable naltrexone; Vivitrol
Behavioral: Motivational Enhancement Therapy and Cognitive Behavioral Therapy — Weekly Motivational Enhancement Therapy and Cognitive Behavioral Therapy (MET/CBT), based upon the Brief Counselling for Marijuana Dependence Manual published by the Substance Abuse and Mental Health Services Administration (SAMHSA), for 12 weeks

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of 12 weeks treatment with an extended-release injectable form of naltrexone (Vivitrol) combined with a psychological intervention in 10 treatment-seeking adults with Cannabis Use Disorder. The hypotheses are that Vivitrol combined with a psychological intervention will be well tolerated, and will reduce cannabis use, improve abstinence rates, and reduce cannabis withdrawal and craving.

DETAILED DESCRIPTION:
This study will be an open-label trial, with no placebo control. Ten male or female treatment-seeking adults with Cannabis Use Disorder (CUD) will be recruited. All participants will receive 3 x 4ml intramuscular injections of Vivitrol (380mg naltrexone). Injections will be administered once every 4 weeks for 12 weeks. In addition, all participants will receive a weekly psychological intervention (Motivational Enhancement Therapy and Cognitive Behavioral Therapy; MET/CBT) for 12 weeks.

The aim of this study is to investigate if the proposed Vivitrol dosing schedule, combined with MET/CBT, is appropriate for subsequent randomized controlled trials in people with CUD. This will be achieved by assessing the safety and effectiveness of 12 weeks open-label treatment with Vivitrol (3 x 4 ml intramuscular injections, 380mg naltrexone) combined with weekly MET/CBT.

Safety will be assessed by monitoring adverse events during the 12 week treatment period, and up to 3 months follow-up. Effectiveness will be assessed after 12 weeks of treatment and at 3 month follow-up using: (1) seven-day point prevalence cannabis abstinence, (2) percentage of days of cannabis use, (3) amount of cannabis use, and (4) effects on withdrawal symptom scores, craving scores and number of urine samples screened positive for cannabis use.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-64) male or female (gender to be analyzed as a covariate)
* Understand and willing to comply with study requirements and restrictions
* Willing to use appropriate contraceptive method throughout the study
* Otherwise healthy as judged by investigator based on medical history, physical exam, vitals, ECG and labs
* DSM 5 criteria for current CUD
* Report cannabis as primary drug of abuse
* Have cannabis positive urine drug screen
* Treatment seeking cannabis smoker

Exclusion Criteria:

* Meets DSM 5 criteria for a current axis I disorder including substance use disorder other than cannabis, nicotine or caffeine dependence.
* Unstable medical conditions
* Pregnant or breast-feeding
* Positive urine drug test for opioids (including methadone, morphine, buprenorphine) or benzodiazepines (unless prescribed) at baseline
* Any IM gluteal administration 30 days prior to baseline
* Participation in a clinical trial of a pharmacological agent within 30 days prior to baseline
* Known intolerance and/or hypersensitivity to naltrexone, carboxymethylcellulose, or polylactide-coglycolide
* Any finding that, in the view of the principal investigator, would compromise the subject's ability to fulfill the protocol visit schedule or visit requirement (e.g. unadjudicated charges and/or pending parole hearings)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD,PhD,MCFP, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vivitrol + MET/CBT
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vivitrol + MET/CBT
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Dropouts Due to Serious Adverse Events
Description: Tolerability will be measured by the number of participants that drop out of the study because of serious adverse events. Adverse events will be monitored weekly during the 12 week treatment phase of the study
Time Frame: At end of 12 weeks treatment
Population: Only 1 participant was enrolled, and this participant withdrew prior to completion at 6 weeks; data are reported up to 6 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Vivitrol + MET/CBT
Number analyzed (Participants) | 1
Participants | 0

2. Primary Outcome: Dropouts Due to Serious Adverse Events
Description: Tolerability will be measured by the number of participants that drop out of the study because of serious adverse events. After the treatment phase of the study adverse events will be monitored weekly for the first 4 weeks follow-up, and then monthly until the final follow-up at 3 months post-treatment
Time Frame: At 3 months follow-up
Population: Only 1 participant was enrolled, and this participant withdrew prior to completion at 6 weeks. Since no participant completed the study and made it to the 3-month follow-up phase, there is no data to report for this outcome.
Arm/Group | Vivitrol + MET/CBT
Number analyzed (Participants) | 0

3. Primary Outcome: Cannabis Abstinence
Description: Seven-day point prevalence of cannabis abstinence. Abstinence will be measured using a self-report timeline follow-back (TLFB) calendar method, and will be confirmed by urine drug screens.
Time Frame: At end of 12 weeks treatment
Population: Only 1 participant was enrolled and this participant withdrew at 6 weeks, so data were not collected for this Outcome Measure.
Arm/Group | Vivitrol + MET/CBT
Number analyzed (Participants) | 0

4. Primary Outcome: Cannabis Abstinence
Description: as for outcome 3
Time Frame: At 3 month follow-up
Population: as for outcome 3
Arm/Group | Vivitrol + MET/CBT
Number analyzed (Participants) | 0

5. Secondary Outcome: Days Cannabis Use
Description: Percentage of days of cannabis use. This will be calculated using a self-report timeline follow-back (TLFB) calendar method
Time Frame: During 12 weeks of treatment and up to 3 month follow-up
Population: as for outcome 1
Measure: Number; unit: Percentage of days/week
Arm/Group | Vivitrol + MET/CBT
Number analyzed (Participants) | 1
Percentage of days/week
  Week 1 | 100
  Week 2 | 28.6
  Week 3 | 0
  Week 4 | 0
  Week 5 | 0
  Week 6 | 0

6. Secondary Outcome: Amount Cannabis Use
Description: Amount of cannabis used (grams per week). The amount of cannabis consumed will be measured using a self-report timeline follow-back (TLFB) calendar method
Time Frame: During 12 weeks of treatment and up to 3 month follow-up
Population: as for outcome 1
Measure: Number; unit: g/week of cannabis
Arm/Group | Vivitrol + MET/CBT
Number analyzed (Participants) | 1
g/week of cannabis
  Week 1 | 14
  Week 2 | 6
  Week 3 | 0
  Week 4 | 0
  Week 5 | 0
  Week 6 | 0

7. Secondary Outcome: Cannabis Withdrawal
Description: Withdrawal symptom scores. Cannabis withdrawal symptoms will be measured using the Marijuana Withdrawal Checklist (MWC). The 16 item MWC indicates severity of withdrawal in the previous 24 hours. Each item is scored 0-4 (where 4=severe) and the scale is summed. The outcome variable is the total score (the sum of each individual item score), which can vary from 0 to 64; higher scores indicate a worse outcome (i.e., more number/severity of withdrawal symptoms).
Time Frame: During 12 weeks of treatment and up to 3 month follow-up
Population: as for outcome 1
Measure: Number; unit: score on a scale
Arm/Group | Vivitrol + MET/CBT
Number analyzed (Participants) | 1
score on a scale
  Week 1 | 4
  Week 2 | 4
  Week 3 | 7
  Week 4 | 13
  Week 5 | 9
  Week 6 | 9

8. Secondary Outcome: Cannabis Craving
Description: Craving symptom scores. Cannabis craving will be measured using the Marijuana Craving Questionnaire (MCQ). The 12-item MCQ assesses craving along 4 dimensions: compulsivity, emotionality, expectancy, and purposefulness. Each subscale is the sum of 3 items from the questionnaire. Each item is rated from 1 (strongly disagree) to 7 (strongly agree). Each subscale can thus vary from 3 to 21, where higher scores represent more craving (worse outcome).
Time Frame: During 12 weeks of treatment and up to 3 month follow-up
Population: as for outcome 1
Measure: Number; unit: score on a scale
Arm/Group | Vivitrol + MET/CBT
Number analyzed (Participants) | 1
score on a scale
  Week 1 Compulsivity | 3
  Week 1 Emotionality | 3
  Week 1 Expectancy | 5
  Week 1 Purposefulness | 3
  Week 2 Compulsivity | 3
  Week 2 Emotionality | 3
  Week 2 Expectancy | 3
  Week 2 Purposefulness | 3
  Week 3 Compulsivity | 3
  Week 3 Emotionality | 3
  Week 3 Expectancy | 3
  Week 3 Purposefulness | 3
  Week 4 Compulsivity | 3
  Week 4 Emotionality | 3
  Week 4 Expectancy | 3
  Week 4 Purposefulness | 3
  Week 5 Compulsivity | 3
  Week 5 Emotionality | 3
  Week 5 Expectancy | 3
  Week 5 Purposefulness | 3
  Week 6 Compulsivity | 3
  Week 6 Emotionality | 3
  Week 6 Expectancy | 3
  Week 6 Purposefulness | 3

9. Secondary Outcome: Urine Cannabis Screens
Description: Number of urine samples positive for cannabis use. Urine samples will be collected to perform THC metabolite analysis
Time Frame: During 12 weeks of treatment and up to 3 month follow-up
Population: as for outcome 1
Measure: Number; unit: Total number of positive urine samples
Arm/Group | Vivitrol + MET/CBT
Number analyzed (Participants) | 1
Total number of positive urine samples | 6

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Use of SAFTEE guidelines to capture AEs at every visit following consent
Arm/Group | Vivitrol + MET/CBT
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivitrol + MET/CBT (N=1)
Nausea (Nervous system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT04139668/Prot_SAP_000.pdf